CLINICAL TRIAL: NCT00094692
Title: An Evaluation of Treatment of Amblyopia in 7 To <18 Year Olds
Brief Title: An Evaluation of Treatment of Amblyopia in Children 7 To <18 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-93; 2U10EY011751 (NIH)
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2007-05

CONDITIONS: Amblyopia
Keywords: Amblyopia; Patching; Spectacles
MeSH Terms: conditions — Amblyopia | interventions — Eyeglasses; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Eye patch
Device: spectacles
Drug: atropine

SUMMARY:
The goals of this study are:

* To determine the response rate of treatment of amblyopia in 7 to <18 year olds.
* To determine the frequency of recurrence of amblyopia in 7 to <18 year olds after discontinuation of amblyopia treatment.

DETAILED DESCRIPTION:
Most eye care practitioners believe that there is an age beyond which attempting to treat amblyopia is futile. It is generally held that the response to treatment is best when it is instituted at an early age and is poor when attempted after eight years of age. There has not been a prospective clinical trial conducted with appropriate rigor that has evaluated the effect of treatment of amblyopia in children aged 7 years or older. Although available data on the efficacy of amblyopia treatment of older children are limited, there is reason to believe from clinical observations and published case series that treatment could have benefit. In a pilot study of patients 10 to <18 years old with amblyopia, we found that 37 percent of 52 patients showed improvement in the amblyopic eye acuity of 2 or more lines after treatment with part-time patching. However, without a concurrent randomized control group, the results are not conclusive. Although the literature and our pilot study provide support that amblyopia can be improved with treatment, neither the response rate to treatment nor the recidivism rate after cessation of treatment can be well defined. Despite the evidence that amblyopia therapy can be effective in older children, many clinicians do not attempt treatment under the assumption that it will be unsuccessful. Therefore, a clinical trial is needed to provide the requisite data to establish clinical practice guidelines for the treatment of amblyopia in older children. In addition to its importance for patient management, the trial's results will meet the demand for cost effectiveness by health maintenance organizations, large employers, and insurers.

The study is a randomized trial comparing patients treated with spectacles only (Control Group) to patients undergoing active treatment (patching, near activities while patching, and atropine for children under the age of 13) in addition to spectacles (Active Treatment Group). It will enroll a minimum of 90 patients in each of the age groups of 7 to <9, 9 to <11, 11 to <13, and 13 to <18 years old. Patients have follow up visits every 6 weeks (up to a maximum of 24 weeks) until they are classified as either responders or nonresponders based on amblyopic eye visual acuity. At the end of the randomized trial:

* Patients who did not respond to treatment end follow up.
* Patients who responded to treatment continue in their respective treatment groups until visual acuity stops improving.

Once there is no further improvement in visual acuity:

* Patients in the Control Group end follow up
* Patients in the Active Treatment Group discontinue active treatment and have follow up visits at 13 weeks, 26 weeks, and 52 weeks timed from treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged 7 to <18 years and have amblyopia associated with strabismus, anisometropia, or both.
* Visual acuity in the amblyopic eye must be 20/40 to 20/400 inclusive and visual acuity in the sound eye must be 20/25 or better.

Exclusion Criteria:

* Patients must not have received amblyopia treatment (other than spectacles) in the past month or more than one month of amblyopia treatment in the last 6 months.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 507
Dates: Start 2002-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement

CONTACTS AND LOCATIONS:
Overall Officials: Richard W. Hertle, M.D., Study Chair — University of Pittsburgh; Mitchell M. Scheiman, O.D., Study Chair — Pennsylvania College of Optometry
Locations (3):
- United States (3):
  - Wilmer Eye Institute, Baltimore, Maryland
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group. A prospective, pilot study of treatment of amblyopia in children 10 to <18 years old. Am J Ophthalmol. 2004 Mar;137(3):581-3. doi: 10.1016/j.ajo.2003.08.043. PMID 15013894
- [Background] Scheiman MM, Hertle RW, Beck RW, Edwards AR, Birch E, Cotter SA, Crouch ER Jr, Cruz OA, Davitt BV, Donahue S, Holmes JM, Lyon DW, Repka MX, Sala NA, Silbert DI, Suh DW, Tamkins SM; Pediatric Eye Disease Investigator Group. Randomized trial of treatment of amblyopia in children aged 7 to 17 years. Arch Ophthalmol. 2005 Apr;123(4):437-47. doi: 10.1001/archopht.123.4.437. PMID 15824215
- [Background] Hertle RW, Scheiman MM, Beck RW, Chandler DL, Bacal DA, Birch E, Chu RH, Holmes JM, Klimek DL, Lee KA, Repka MX, Weakley DR Jr; Pediatric Eye Disease Investigator Group. Stability of visual acuity improvement following discontinuation of amblyopia treatment in children aged 7 to 12 years. Arch Ophthalmol. 2007 May;125(5):655-9. doi: 10.1001/archopht.125.5.655. PMID 17502505
- [Derived] Wallace DK, Lazar EL, Melia M, Birch EE, Holmes JM, Hopkins KB, Kraker RT, Kulp MT, Pang Y, Repka MX, Tamkins SM, Weise KK; Pediatric Eye Disease Investigator Group. Stereoacuity in children with anisometropic amblyopia. J AAPOS. 2011 Oct;15(5):455-61. doi: 10.1016/j.jaapos.2011.06.007. PMID 22108357
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898